CLINICAL TRIAL: NCT03969459
Title: Impact of Exposure to Persistent Organic Pollutants During Pregnancy on the Composition of Breast Milk and Consequences on the Newborn
Acronym: PESTIMICOBLAIT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0032
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Pesticide; Breast Milk; Pollution; Exposure; Meconium; Stool; Microbiota; Newborn
Keywords: pesticide exposure; persistent organic pollutants; breast milk; meconium; stool; microbiota; newborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast milk for the mother, meconium and feces for the newborn
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: breast milk collection — 3 samples of 20 ml of breast milk will be collected between day 0 and day 4; between day 7 and day 15; and between day 21 and day 30 after childbirth.
Biological: meconium collection — 3 samples of 20 ml of meconium milk will be collected between day 0 and day 4; between day 7 and day 15; and between day 21 and day 30 after childbirth.
Biological: newborn feces collection — 3 samples of 20 ml of newborn feces will be collected between day 0 and day 4; between day 7 and day 15; and between day 21 and day 30 after childbirth.
Other: questionary of pesticide exposure of the mother — maternal questionary of pesticide exposure of the mother

SUMMARY:
Epidemiological studies link early exposure to persistent organic pollutants (POPs) with health consequences in the newborn. Experimental studies have shown the impact of POPs on the gut microbiota. This project aims to characterize the POPs content in breast milk in an exposed population and to evaluate the impact on breast milk composition and intestinal microbiota establishment in the newborn. The health consequences will be evaluated by the clinical follow-up of the newborn.

DETAILED DESCRIPTION:
Picardie is a sub-region with a young population and a high birth rate. The highlighting and the characterization of a maternal exhibition and the newborn will make it possible to know the in utero and postnatal exposure to the pesticides, and if necessary, to implement measures of information and prevention adapted to limit it.

The study of pesticide exposure in the periconceptional period, ante and postnatal is crucial because of the vulnerability of this period to the environment and its immediate consequences on the health of the child but also in the long term on the development of chronic pathologies in adulthood. This study will allow us to assess the impact of POPs on the installation of the intestinal microbiota of newborn.

100 mother-child pairs will be included in this project. Samples of 20 mL of breast milk, meconium and stool of newborns will be taken. Gas chromatography or liquid phase analyzes coupled with mass spectrometry will be carried out on breast milk to evaluate the content of persistent organic pollutants and to isolate them. An analysis of the chemical composition of each milk sample will be performed. A bacteriological study for the enumeration of the germs in the mother's milk on the one hand then in the meconium and the saddles of the new-born on the other part will be realized. The DNA of isolated and identified germs will be compared by molecular biology techniques to determine their identity or non-identity within the microbiota of breast milk, meconium and newborn stool. The impact of breast milk contamination by pesticides on the health of newborn will be studied

ELIGIBILITY:
Inclusion Criteria:

* newborn born before 33 weeks of amenorrhea or at term born at least 37 weeks of amenorrhea
* mother aged of 18 to 42 years old at the time of inclusion
* mother not deprived of parental rights
* signed concerned consent
* mother having lived for at least 6 months in the Picardie subregion

Exclusion Criteria:

* newborn whose term of birth is between 33 and 37 weeks of amenorrhea
* mother minor or aged over 42 years
* mother deprived of her parental rights

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 100 mother-child pairs will be included in this project Newborn were born before 33 weeks of amenorrhea or at term born at least 37 weeks of amenorrhea.
  mother are aged of 18 to 42 years old at the time of inclusion
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
measure of quantity of pesticides in mother's milk | between day 0 and day 4 after childbirth
  the evaluation of the contamination of the mother's milk by pesticides will be done on 20 ml sample of breast milk.
measure of quantity of pesticides in mother's milk | between day 7 and day 15 after childbirth
  the evaluation of the contamination of the mother's milk by pesticides will be done on 20 ml sample of breast milk.
measure of quantity of pesticides in mother's milk | between day 21 and day 30 after childbirth
  the evaluation of the contamination of the mother's milk by pesticides will be done on 20 ml sample of breast milk.

SECONDARY OUTCOMES:
correlation between measure of quantity of pesticides in mother's milk and microbiota composition in mother's milk | between day 0 and day 4 after childbirth
  correlation between pesticides contamination of mother's milk and microbiota composition in mother's milk
correlation between measure of quantity of pesticides in mother's milk and microbiota composition in mother's milk | between day 7 and day 15 after childbirth
  correlation between pesticides contamination of mother's milk and microbiota composition in mother's milk
correlation between measure of quantity of pesticides in mother's milk and microbiota composition in mother's milk | between day 21 and day 30 after childbirth
  correlation between pesticides contamination of mother's milk and microbiota composition in mother's milk

CONTACTS AND LOCATIONS:
Overall Officials: Andre Leke, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No